CLINICAL TRIAL: NCT02970643
Title: Proof-of-Concept Trial of Palonosetron and Olanzapine Without Dexamethasone for the Prevention of Chemotherapy-Induced Nausea and Vomiting
Brief Title: Proof-of-Concept Trial of Palonosetron and Olanzapine Without Dexamethasone for the Prevention of CIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hee Jun Kim (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Sponsor-Investigator, Hee Jun Kim, Associate Professor,Division of Hemato-oncology, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Organization: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C2016034
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Olanzapine; Chemotherapy-Induced Nausea and Vomiting; Moderate risk
MeSH Terms: conditions — Vomiting | interventions — Olanzapine; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olanzapine group (Experimental): Palonosetron and Olanzapine Without Dexamethasone in moderate risk chemotherapy induced nausea and vomiting group
  Interventions: Drug: Olanzapine; Drug: Palonosetron

INTERVENTIONS:
Drug: Olanzapine — Moderate risk chemotherapy induced nausea group in all cancer. D1 Olanzapine 10mg PO D2-3 Olanzapine 10mg PO
  Other Names: Zyprexa
Drug: Palonosetron — Moderate risk chemotherapy induced nausea group in all cancer. D1 Palonosetron 0.25mg IV
  Other Names: Aloxi

SUMMARY:
The purpose of this study is to determine whether Palonosetron and Olanzapine without dexamethasone for the Prevention of moderate risk Chemotherapy-Induced Nausea and vomiting.

DETAILED DESCRIPTION:
This study was designed to evaluate efficacy and safety of olanzapine compared with 5-hydroxytryptamine3 receptor antagonist for prevention of moderate risk chemotherapy induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* European Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* no severe cognitive compromise
* Moderate risk chemotherapy induced chemotherapy induced nausea and vomiting in 1st cycle
* Confirmed histology

Exclusion Criteria:

* European Cooperative Oncology Group (ECOG) performance status of 3 and 4
* Nausea or vomiting in the 24 hours before enrollment
* History of Nausea or vomiting Grade 3 before previous chemotherapy
* Known history of central nervous system disease (e.g., brain metastases or a seizure disorder)
* Bowel obstruction
* Serum creatinine level of 2.0 mg per deciliter (177 μmol per liter) or more
* Aspartate or alanine aminotransferase level that was more than 3 times the upper limit of the normal range
* Treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, a phenothiazine, or a butyrophenone within 30 days before enrollment
* Treatment with another antiemetic agent before 48 hours before enrollment
* Uncontrolled severe infection or uncontrolled severe comorbidity
* Concurrent abdominal radiotherapy
* Known hypersensitivity to olanzapine, palonosetron
* Known cardiac arrhythmia, uncontrolled congestive heart failure, or acute myocardial infarction within the previous 6 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 4.0 nausea | the overall assessment period (0 to 72 hours)

SECONDARY OUTCOMES:
Quality of life was evaluated according to MDASI-K | the overall assessment period (0 to 72 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Heejun Kim, MD.PhD, Study Chair — Associate Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navari RM, Qin R, Ruddy KJ, Liu H, Powell SF, Bajaj M, Dietrich L, Biggs D, Lafky JM, Loprinzi CL. Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Jul 14;375(2):134-42. doi: 10.1056/NEJMoa1515725. PMID 27410922
- [Background] Tan L, Liu J, Liu X, Chen J, Yan Z, Yang H, Zhang D. Clinical research of Olanzapine for prevention of chemotherapy-induced nausea and vomiting. J Exp Clin Cancer Res. 2009 Sep 23;28(1):131. doi: 10.1186/1756-9966-28-131. PMID 19775450
- [Background] Naeim A, Dy SM, Lorenz KA, Sanati H, Walling A, Asch SM. Evidence-based recommendations for cancer nausea and vomiting. J Clin Oncol. 2008 Aug 10;26(23):3903-10. doi: 10.1200/JCO.2007.15.9533. PMID 18688059
- [Background] Lohr L. Chemotherapy-induced nausea and vomiting. Cancer J. 2008 Mar-Apr;14(2):85-93. doi: 10.1097/PPO.0b013e31816a0f07. PMID 18391612
- [Background] American Society of Clinical Oncology; Kris MG, Hesketh PJ, Somerfield MR, Feyer P, Clark-Snow R, Koeller JM, Morrow GR, Chinnery LW, Chesney MJ, Gralla RJ, Grunberg SM. American Society of Clinical Oncology guideline for antiemetics in oncology: update 2006. J Clin Oncol. 2006 Jun 20;24(18):2932-47. doi: 10.1200/JCO.2006.06.9591. Epub 2006 May 22. PMID 16717289
- [Background] Navari RM, Gray SE, Kerr AC. Olanzapine versus aprepitant for the prevention of chemotherapy-induced nausea and vomiting: a randomized phase III trial. J Support Oncol. 2011 Sep-Oct;9(5):188-95. doi: 10.1016/j.suponc.2011.05.002. Epub 2011 Sep 24. PMID 22024310
- [Background] Vardy J, Chiew KS, Galica J, Pond GR, Tannock IF. Side effects associated with the use of dexamethasone for prophylaxis of delayed emesis after moderately emetogenic chemotherapy. Br J Cancer. 2006 Apr 10;94(7):1011-5. doi: 10.1038/sj.bjc.6603048. PMID 16552437
- [Background] Cleeland CS, Mendoza TR, Wang XS, Chou C, Harle MT, Morrissey M, Engstrom MC. Assessing symptom distress in cancer patients: the M.D. Anderson Symptom Inventory. Cancer. 2000 Oct 1;89(7):1634-46. doi: 10.1002/1097-0142(20001001)89:73.0.co;2-v. PMID 11013380